CLINICAL TRIAL: NCT01732484
Title: Posterior Capsule Opacification and Frequency of Nd:YAG Treatment and of Two Microincision IOLs: Hoya iMics NY-60 vs Acrysof SN60WF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Prof. Dr. Rupert Menapace, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: EK1444/2012
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Results first posted 2013-06-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-04

CONDITIONS: Capsule Opacification; Pseudophakia; Cataract
MeSH Terms: conditions — Capsule Opacification; Pseudophakia; Cataract | interventions — Lens Implantation, Intraocular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- iMics1 NY-60 (Other): eyes with implantation of iMics1 NY-60 IOL
  Interventions: Procedure: intraocular lens implantation
- AcrySof SN60WF (Other): eyes with implantation of AcrySof SN60WF IOL
  Interventions: Procedure: intraocular lens implantation

INTERVENTIONS:
Procedure: intraocular lens implantation

SUMMARY:
Age-related cataract is the main cause of impaired vision in the elderly population worldwide. In the UK, more than half of people who are over 65 have some cataract development in one or both eyes. The only treatment that can restore functional visual ability is cataract surgery where the opacified crystalline lens is removed by phacoemulsification and an artificial intraocular lens is implanted. It is estimated that around 10 million cataract operations are performed around the world each year. Cataract operations are generally very successful, with a low risk of serious complications. The most common risk is developing a condition called posterior capsule opacification (PCO), which causes impaired vision to return.

During the past two decades, cataract surgery underwent tremendous change and modernisation resulting in today's small incision phacoemulsification surgery and a safe technique with a short rehabilitation time for the patient. The most frequent long-term complication of cataract surgery remains to be posterior capsule opacification (PCO). In the past few years, refinements in surgical technique and modifications in IOL design and material have led to a decrease in the incidence of PCO.

It has been shown that a sharp posterior optic edge inhibits migration of lens epithelial cells (LEC) behind the IOL optic and therefore have a lower incidence of posterior capsule opacification (PCO). Most IOL designs have open-loop haptics that are connected to the optic towards the end of the production process, also called multipiece designs.

For several reasons such as better ease of use with injector systems and higher efficiency in the production process, companies have developed IOLs with open-loop haptics out of one block of material, also called single-piece designs. In the case of such single-piece IOLs, the haptics tend to be much thicker than with multipiece IOLs. A potential drawback of the thick haptics maybe an incomplete closure of the capsule at the optic rim with a reduced bending effect of the posterior capsule around the posterior optic edge. Additionally, the posterior sharp edge is often discontinuous in the region of the haptic-optic junctions. These locations may serve as a scaffold for LECs to migrate behind the IOL optic resulting in PCO. Nowadays a multitude of different single piece IOLS are available, many of them similar but of course with some differences in regard to the chemical composition of the acrylic material and the IOL design.

The purpose of this study is to compare the intensity of posterior capsule opacification (PCO) between two different 1-piece foldable hydrophobic acrylic intraocular lenses (IOLs) over a period of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* bilateral age-related cataract
* good overall physical constitution

Exclusion Criteria:

* history of ocular disease or intraocular surgery
* laser treatment
* diabetes requiring medical control
* glaucoma
* severe retinal pathology that would make a postoperative visual acuity of 20/40 (decimal equivalent = 0.5) or better unlikely

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Menapace, MD, Principal Investigator — Medical University Vienna

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Included
Started | 100
Randomized | 100 (Randomized implantation SN60WF IOL in on eye and iMics NY-60 in the other eye.)
Allocation | 100
Completed | 74
Not Completed | 26
Not completed — Death | 7
Not completed — Lost to Follow-up | 14
Not completed — chronical illness | 5

BASELINE CHARACTERISTICS:
Groups:
- Cataract Surgery: eyes with implantation of iMics1 NY-60 IOL or Acrysof SN60WF IOL
Arm/Group | Cataract Surgery
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 100
Age Continuous [Mean (Standard Deviation); unit: years] | 72 (9)
Gender [Number; unit: participants]
  Female | 42
  Male | 32
Region of Enrollment [Number; unit: participants]
  Austria | 100

OUTCOME MEASURES:

1. Primary Outcome: Posterior Capsule Opacification (PCO)
Description: PCO = migration of lens epithelial cells behind the IOL optic after cataract surgery; scale 0-10 (0: no PCO; 10: maximum PCO)
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: units on a scale (0-10)
Arm/Group | iMics1 NY-60 | AcrySof SN60WF
Number analyzed (Participants) | 74 | 74
units on a scale (0-10) | 3.0 (2.0) | 1.9 (1.4)

2. Secondary Outcome: Percentage of Eyes With Neodymium:Yttrium-aluminium-garnet (Nd:YAG) Capsulotomy
Description: Treatment of PCO in neodymium:yttrium-aluminium-garnet (Nd:YAG) capsulotomy. The frequency of this treatment will be asseseed in percentage values
Time Frame: 3 years
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | iMics1 NY-60 | AcrySof SN60WF
Number analyzed (Participants) | 74 | 74
Number analyzed (eyes) | 148 | 148
percentage of eyes | 26 (0) | 10 (0)

ADVERSE EVENTS:
Arm/Group | iMics1 NY-60 | AcrySof SN60WF
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes